CLINICAL TRIAL: NCT04568811
Title: The Single-center, Open-label Phase I Clinical Trial of Booster Vaccination of Adenovirus Type-5 Vectored COVID-19 Vaccine in Healthy Adults Aged 18-60 Years
Brief Title: The Phase I Clinical Trial of Booster Vaccination of Adenovirus Type-5 Vectored COVID-19 Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: JSVCT100
Record Dates: First submitted 2020-09-28; First posted 2020-09-29 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Adenovirus Type-5 Vectored COVID-19 Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adenovirus Type-5 Vectored COVID-19 Vaccine (Experimental)
  Interventions: Biological: Adenovirus Type-5 Vectored COVID-19 Vaccine

INTERVENTIONS:
Biological: Adenovirus Type-5 Vectored COVID-19 Vaccine — Low dose adenovirus type-5 vectored COVID-19 vaccine (5E10 vp)

SUMMARY:
The 2019 novel-coronavirus (2019-nCov) is the cause of a cluster of unexplained pneumonia that started in Hubei province in China. It has manifest into a global health crisis with escalating confirmed cases and spread across many countries.

In view of the fact that there is currently no effective antiviral therapy, the prevention or treatment of diseases caused by COVID-19 can be tough for current treatment.

This study is a phase I clinical trial of booster vaccination of adenovirus type-5 vectored COVID-19 vaccine 6 months after prime vaccination. The investigators intent to evaluate the safety and immunogenicity of booster vaccination of adenovirus type-5 vectored COVID-19 vaccine in healthy adults aged aged 18-60 years.

DETAILED DESCRIPTION:
The 2019 novel-coronavirus (2019-nCov) is the cause of a cluster of unexplained pneumonia that started in Hubei province in China. It has manifest into a global health crisis with escalating confirmed cases and spread across many countries.

In view of the fact that there is currently no effective antiviral therapy, the prevention or treatment of diseases caused by COVID-19 can be tough for current treatment.

This is a single-center, open-label phase I clinical trial of booster vaccination in healthy 18 to 60 years of age, inclusive, who has been prime vaccinated with adenovirus type-5 vectored COVID-19 vaccine. This clinical trial is designed to assess the safety and immunogenicity of booted vaccination of adenovirus type-5 vectored COVID-19 vaccine manufactured by Beijing Institute of Biotechnology and CanSino Biologics Inc.

ELIGIBILITY:
Inclusion Criteria:

* Participants who has received prime vaccination of adenovirus type-5 vectored COVID-19 vaccine
* Able to understand the content of informed consent and willing to sign the informed consent
* Negative in HIV diagnostic test.
* Axillary temperature ≤37.0°C.
* General good health as established by medical history and physical examination.
* Able to complete 12 months visit

Exclusion Criteria:

* Family history of seizure, epilepsy, brain or mental disease
* Subject allergic to any component of the investigational vaccine, or a more severe allergic reaction and history of allergies in the past.
* Woman who is pregnant, breast-feeding on day of enrollment, or become pregnant during the next 12 months
* Any acute fever disease or infections.
* History of SARS
* Major congenital defects or not well-controlled chronic illness, such as asthma, diabetes, or thyroid disease.
* Serious cardiovascular diseases, such as arrhythmia, conduction block, myocardial infarction, severe hypertension without controllable drugs, etc.
* Hereditary angioneurotic edema or acquired angioneurotic edema
* Urticaria in last one year
* No spleen or functional spleen.
* Platelet disorder or other bleeding disorder may cause injection contraindication
* Faint at the sight of needles.
* Prior administration of immunodepressant or corticosteroids, antianaphylaxis treatment, cytotoxic treatment in last 6 months.
* Prior administration of blood products in last 4 months
* Prior administration of other research medicines in last 1 month
* Prior administration of attenuated vaccine in last 1 month
* Prior administration of inactivated vaccine in last 14 days
* Current anti-tuberculosis prophylaxis or therapy
* According to the judgement of investigator,various medical, psychological, social or other conditions, those could affect the subjects to sign informed consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2020-09-26 (Actual); Primary Completion 2020-10-25 (Actual); Study Completion 2021-09-11 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse reactions within 14 days after booster vaccination | 0-14 days post-vaccination
  Occurrence of adverse reactions within 14 days after booster vaccination of adenovirus type-5 vectored COVID-19 vaccine

SECONDARY OUTCOMES:
Occurrence of adverse events within 14 days after booster vaccination | 0-14 days post-vaccination
  Occurrence of adverse events within 14 days after booster vaccination of adenovirus type-5 vectored COVID-19 vaccine
Occurrence of adverse events within 28 days after booster vaccination | 0-28 days post-vaccination
  Occurrence of adverse events within 28 days after booster vaccination of adenovirus type-5 vectored COVID-19 vaccine
Occurrence of serious adverse events within 28 days after booster vaccination | 0-28 days post-vaccination
  Occurrence of serious adverse events within 28 days after booster vaccination of adenovirus type-5 vectored COVID-19 vaccine
Occurrence of serious adverse events within 6 months after booster vaccination | 6 months post-vaccination
  Occurrence of serious adverse events within 6 months after booster vaccination of adenovirus type-5 vectored COVID-19 vaccine
Occurrence of serious adverse events within 12 months after booster vaccination | 12 months post-vaccination
  Occurrence of serious adverse events within 12 months after booster vaccination of adenovirus type-5 vectored COVID-19 vaccine
Changes in laboratory test indicators before and 1 day after vaccination | 1 day post-vaccination
  Changes in laboratory test indicators (including white blood cell count, lymphocyte count, neutrophils, platelets, hemoglobin, ALT, AST, total bilirubin, fasting blood glucose, creatinine) before and 1 day after vaccination
Antibody of S-RBD at day 14, day 28, month 6 and month 12 after booster vaccination | 14 days, 28 days, 6 months and 12 months post-vaccination
  Antibody of S-RBD at day 14, day 28, month 6 and month 12 after booster vaccination of adenovirus type-5 vectored COVID-19 vaccine
Cellular immunity at day 14 after booster vaccination | 14 days post-vaccination
  Cellular immunity at day 14 after booster vaccination of adenovirus type-5 vectored COVID-19 vaccine

CONTACTS AND LOCATIONS:
Locations (1):
- A rehabilitation centre in Wuhan, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jia S, Zhang J, Wang X, Zhang Z, Wang B, Zhang J, Jiang H, Guo G, Wang Y, Wan J, Wang W, Hou L, Zhu F. Safety and Immunogenicity of Homologous Recombinant Adenovirus Type 5-Vectored COVID-19 Vaccine Booster Dose in Healthy Adults Aged 18-60 Years: a Single-Center, Open-Label Trial. Infect Dis Ther. 2023 Dec;12(12):2757-2769. doi: 10.1007/s40121-023-00892-0. Epub 2023 Dec 1. PMID 38038866